CLINICAL TRIAL: NCT03326674
Title: A Multinational, Multicenter, Randomized, Phase 3 Study of Tesetaxel Plus a Reduced Dose of Capecitabine Versus Capecitabine Alone in Patients With HER2 Negative, HR Positive, Locally Advanced or Metastatic Breast Cancer Previously Treated With a Taxane
Brief Title: Tesetaxel Plus Reduced Dose of Capecitabine vs. Capecitabine in HER2 Negative, HR Positive, LA/MBC
Acronym: CONTESSA
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The Sponsor has discontinued the development of tesetaxel
Sponsor: Odonate Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ODO-TE-B301
Record Dates: First submitted 2017-10-13; First posted 2017-10-31 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Breast Cancer
Keywords: Tesetaxel; Capecitabine; HER2 negative; Hormone Receptor positive; Locally advanced or metastatic breast cancer; Combination of tesetaxel and capecitabine; Taxanes; Metastatic breast cancer; Breast cancer; Central nervous system (CNS) metastases
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — tesetaxel; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Tesetaxel (oral) and capecitabine (oral) (Experimental): Tesetaxel (27 mg/m2) once every 21 days on Day 1 of each 21-day cycle; and capecitabine (825 mg/m2) twice daily (in the morning and evening after a meal, for a total daily dose of 1,650 mg/m2) beginning with the evening dose on Day 1 through the morning dose on Day 15 of each 21-day cycle
  Interventions: Drug: Tesetaxel and Capecitabine
- Arm B: Capecitabine (oral) (Active Comparator): Capecitabine (1,250 mg/m2) twice daily (in the morning and evening after a meal, for a total daily dose of 2,500 mg/m2) beginning with the evening dose on Day 1 through the morning dose on Day 15 of each 21-day cycle
  Interventions: Drug: Capecitabine

INTERVENTIONS:
Drug: Tesetaxel and Capecitabine — Tesetaxel plus reduced dose of Capecitabine
  Arms: Arm A: Tesetaxel (oral) and capecitabine (oral)
Drug: Capecitabine — Capecitabine alone at approved dose
  Arms: Arm B: Capecitabine (oral)

SUMMARY:
CONTESSA is a multinational, multicenter, randomized, Phase 3 study of tesetaxel in patients with HER2 negative, HR positive LA/MBC previously treated with a taxane in the neoadjuvant or adjuvant setting. The primary objective of the study is to compare the efficacy of tesetaxel plus a reduced dose of capecitabine versus the approved dose of capecitabine alone based on progression-free survival (PFS) as assessed by the Independent Radiologic Review Committee (IRC). 685 patients were enrolled.

DETAILED DESCRIPTION:
CONTESSA is a multinational, multicenter, randomized, Phase 3 study of tesetaxel plus a reduced dose of capecitabine versus the approved dose of capecitabine alone in patients with HER2 negative, HR positive locally advanced or metastatic breast cancer (LA/MBC) previously treated with a taxane in the neoadjuvant or adjuvant setting. 685 patients were enrolled, including 674 who received treatment.

Patients randomly assigned to Arm A (tesetaxel plus a reduced dose of capecitabine) are administered:

* Tesetaxel (27 mg/m2) orally once every 21 days on Day 1 of each 21-day cycle; and
* Capecitabine (825 mg/m2) orally twice daily (in the morning and evening after a meal, for a total daily dose of 1,650 mg/m2) beginning with the evening dose on Day 1 through the morning dose on Day 15 of each 21-day cycle.

Patients randomly assigned to Arm B (approved dose of capecitabine alone) are administered:

* Capecitabine (1,250 mg/m2) orally twice daily (in the morning and evening after a meal, for a total daily dose of 2,500 mg/m2) beginning with the evening dose on Day 1 through the morning dose on Day 15 of each 21-day cycle

Dose modifications for tesetaxel and/or capecitabine are described in the study protocol.

Patients are treated until documentation of progressive disease (PD), evidence of unacceptable toxicity or other decision to discontinue treatment. Capecitabine is an oral chemotherapy agent that is considered a standard-of-care treatment in LA/MBC. The primary efficacy endpoint is PFS as assessed by the IRC. The secondary efficacy endpoints are overall survival (OS), objective response rate (ORR) as assessed by the IRC and disease control rate (DCR) as assessed by the IRC.

ELIGIBILITY:
Inclusion Criteria:

1. Female or male patients at least 18 years of age
2. Histologically or cytologically confirmed breast cancer
3. HER2 negative disease based on local testing: American Society of Clinical Oncology/College of American Pathologists (ASCO/CAP) guidelines should be utilized for assessing HER2 status
4. HR (estrogen receptor [ER] and/or progesterone receptor [PgR]) positive disease based on local testing: ASCO/CAP guidelines should be utilized for assessing HR status
5. Measurable disease per RECIST 1.1 or bone-only disease with lytic component

   * Patients with bone-only metastatic cancer must have a lytic or mixed lytic-blastic lesion that can be accurately assessed by computerized tomography (CT) or magnetic resonance imaging (MRI). Patients with bone-only disease without a lytic component (ie, blastic-only metastasis) are not eligible.
   * Known metastases to the CNS are permitted but not required. The following criteria apply:

     * Patients must be neurologically stable and either off corticosteroids or currently treated with a maximum daily dose of 4 mg of dexamethasone (or equivalent), with no increase in corticosteroid dose within 7 days prior to randomization
     * Patients with a history of CNS metastases but with no current evidence of CNS lesions following local therapy are eligible
     * Patients may have CNS metastases that are stable or progressing radiologically
     * Patients with current evidence of leptomeningeal disease are not eligible
     * Patients may have untreated brain metastases or previously treated brain metastases, as long as no immediate local CNS-directed therapy is indicated
     * Any prior whole brain radiation therapy must have been completed > 14 days prior to the date of randomization
     * Prior stereotactic brain radiosurgery is permitted
     * CNS surgical resection must have been completed > 28 days prior to the date of randomization; patient must have complete recovery from surgery
6. Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, or 2
7. Prior therapy (at least one completed dose) with a taxane-containing regimen in the neoadjuvant or adjuvant setting
8. Prior therapy with an anthracycline-containing regimen in the neoadjuvant, adjuvant, or metastatic setting, where indicated by local regulation or Investigator judgment.
9. Prior endocrine therapy with or without a CDK 4/6 inhibitor unless endocrine therapy is not indicated (ie, short relapse-free interval while on adjuvant endocrine therapy [endocrine resistance]; rapidly progressing disease/visceral crisis; or endocrine intolerance). Any targeted therapies approved for HER2 negative, HR positive LA/MBC, including everolimus, are permitted as prior therapy. There is no limit to the number of prior endocrine therapies.
10. Documented disease recurrence or disease progression of: (a) locally advanced disease that is not considered curable by surgery and/or radiation; or (b) metastatic disease.
11. Adequate hematologic, hepatic and renal function, as evidenced by:

    * Absolute neutrophil count (ANC) ≥ 1,500/μL without colony-stimulating factor support
    * Platelet count ≥ 100,000/μL
    * Hemoglobin ≥ 10 g/dL without need for hematopoietic growth factor or transfusion support
    * Total bilirubin < 1.5 × upper limit of normal (ULN); does not apply to patients with Gilbert's syndrome
    * Alanine aminotransferase (ALT) < 3 × ULN unless hepatic metastases are present, then < 5 × ULN
    * Aspartate aminotransferase (AST) < 3 × ULN unless hepatic metastases are present, then < 5 × ULN
    * Alkaline phosphatase < 2.5 × ULN unless hepatic metastases are present, then < 5 × ULN
    * Calculated creatinine clearance ≥ 50 mL/min (by Cockcroft-Gault formula or local standard)
    * Serum albumin ≥ 3.0 g/dL
    * Prothrombin time (PT) < 1.5 × ULN or international normalized ratio (INR) < 1.3, and partial thromboplastin time (PTT) < 1.5 × ULN, unless the patient is on a therapeutic anticoagulant
12. Complete recovery to baseline or Grade 1 per National Cancer Institute (NCI) CTCAE version 5.0 from adverse effects of prior surgery, radiotherapy, endocrine therapy and other therapy, as applicable, with the exception of Grade 2 alopecia from prior chemotherapy
13. Ability to swallow an oral solid-dosage form of medication
14. A negative serum pregnancy test within 7 days prior to the first dose of Study treatment in women of childbearing potential (ie, all women except those who are post menopause for ≥ 1 year or who have a history of hysterectomy or surgical sterilization)
15. Women of childbearing potential must use an effective, non-hormonal form of contraception from Screening throughout the Treatment Phase and until 70 days after the last dose of study treatment

    • Acceptable methods include: copper intrauterine devices or double barrier methods, including male/female condoms with spermicide and use of contraceptive sponge, cervical cap, or diaphragm
16. Male patients must use an effective, non-hormonal form of contraception from screening throughout the treatment phase and until 130 days after last dose of study treatment

    • Acceptable methods include male/female condoms with spermicide, or vasectomy with medical confirmation of surgical success
17. Written informed consent and authorization to use and disclose health information
18. Ability to comprehend and comply with the requirements of the study

Exclusion Criteria:

1. Two or more prior chemotherapy regimens for advanced disease
2. Prior treatment with a taxane in the metastatic setting
3. Prior treatment with capecitabine at any dose
4. Current evidence of leptomeningeal disease
5. Other cancer that required therapy within the preceding 5 years other than adequately treated: (a) non-melanoma skin cancer or in situ cancer; or (b) following approval by the Medical Monitor, other cancer that has a very low risk of interfering with the safety or efficacy endpoints of the study
6. Known human immunodeficiency virus infection, unless well controlled. Patients who are on an adequate antiviral regimen with no evidence of active infection are considered well controlled.
7. Active hepatitis B or active hepatitis C infection
8. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the patient inappropriate for entry into this study
9. Presence of neuropathy > Grade 1 per NCI CTCAE version 5.0
10. History of hypersensitivity to taxanes; hypersensitivity to the solvent does not preclude patient participation in this study
11. Anticancer treatment, including endocrine therapy, radiotherapy (except stereotactic brain radiosurgery), chemotherapy, biologic therapy, or therapy in an investigational clinical study, ≤ 14 days prior to the date of randomization
12. Major surgery ≤ 28 days prior to the date of randomization; patient must have complete recovery from surgery
13. Less than 2 weeks or 5 plasma half-lives (whichever is greater) since last use of a medication or ingestion of an agent, beverage or food that is a known clinically relevant strong inhibitor or known clinically relevant inducer of the cytochrome P450 (CYP) 3A pathway (patients should discontinue taking any regularly taken medication that is a strong inhibitor or inducer of the CYP3A pathway)
14. History of hypersensitivity or unexpected reactions to capecitabine, other fluoropyrimidine agents or any of their ingredients
15. Known dihydropyrimidine dehydrogenase (DPD) deficiency. Testing for DPD deficiency must be performed where required by local regulations, using a validated method that is approved by local health authorities.
16. Pregnant or breastfeeding
17. If, in the opinion of the Investigator, the patient is deemed unwilling or unable to comply with the requirements of the study
18. Treatment with brivudine, sorivudine or its chemically-related analogs ≤ 28 days prior to the date of randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 685 (Actual)
Dates: Start 2017-12-21 (Actual); Primary Completion 2020-08-24 (Actual); Study Completion 2021-06-28 (Actual)

PRIMARY OUTCOMES:
PFS as assessed by the IRC | Approximately 2.5-3.0 years

SECONDARY OUTCOMES:
OS | Approximately 5.0-5.5 years
ORR as assessed by the IRC | Approximately 2.5-3.0 years
DCR as assessed by the IRC | Approximately 2.5-3.0 years
Central nervous system (CNS) ORR as assessed by the CNS IRC in patients with CNS metastases at baseline | Approximately 2.5-3.0 years
CNS PFS as assessed by the CNS IRC in patients with CNS metastases at baseline or a history of CNS metastases and in the intent-to-treat (ITT) population | Approximately 2.5-3.0 years
CNS OS in patients with CNS metastases at baseline or a history of CNS metastases | Approximately 2.5-3.0 years

OTHER OUTCOMES:
European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-C30 (EORTC QLQ-C30) Global Health Status/QoL | Approximately 2.5-3.0 years
EORTC QLQ-C30 Functional Scales and Symptom Scales/Items | Approximately 2.5-3.0 years
Adverse events, including deaths and other serious adverse events | Approximately 5.0-5.5 years
Incidence of clinical laboratory abnormalities (e.g., CBC, serum chemistry and coagulation testing) | Approximately 5.0-5.5 years
Peak plasma concentration (Cmax) of tesetaxel | Approximately 2.5-3.0 years
Area under the plasma concentration versus time curve (AUC) of tesetaxel | Approximately 2.5-3.0 years

CONTACTS AND LOCATIONS:
Overall Officials: Joseph O'Connell, MD, Study Director — Odonate Therapeutics, Inc.
Locations (207):
- United States (90):
  - Ironwood Cancer and Research Centers, Chandler, Arizona
  - Cancer Treatment Centers of America - Western Regional Medical Center, Goodyear, Arizona
  - Arizona Oncology Associates, P.C. - HOPE, Tucson, Arizona
  - Genesis Cancer Center, Hot Springs, Arkansas
  - Carti Cancer Center, Little Rock, Arkansas
  - Pacific Cancer Medical Center, Anaheim, California
  - CBCC Global Research, Inc., Bakersfield, California
  - Compassionate Care Research Group, Fountain Valley, California
  - California Cancer Associates for Research and Excellence, Fresno, California
  - St. Joseph Heritage Healthcare, Fullerton, California
  - UCLA Medical Center, Los Angeles, California
  - Cancer Care - Torrance Memorial Physician Network, Redondo Beach, California
  - Sharp Memorial Hospital, San Diego, California
  - University of California San Francisco - Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - San Luis Obispo Oncology & Hematology Health Center, San Luis Obispo, California
  - California Cancer Associates for Research and Excellence, San Marcos, California
  - Cancer Research Collaboration and Breast Link, Santa Ana, California
  - Stanford Cancer Center / Cancer Clinical Trials, Stanford, California
  - Innovative Clinical Research Institute, Whittier, California
  - Rocky Mountain Cancer Center, Lakewood, Colorado
  - Western Connecticut Health Network, Danbury, Connecticut
  - Hartford Healthcare, Hartford, Connecticut
  - Sarah Cannon Research Institute - Florida Cancer Specialists, Fort Myers, Florida
  - Memorial Healthcare System, Hollywood, Florida
  - Cancer Specialists of North Florida, Jacksonville, Florida
  - Miami Cancer Institute, Miami, Florida
  - Florida Cancer Affiliates - Ocala, Ocala, Florida
  - Orlando Health, Orlando, Florida
  - University of Miami Sylvester Comprehensive Cancer Center / Sylvester at Plantation, Plantation, Florida
  - Florida Cancer Specialists and Research Institute, St. Petersburg, Florida
  - Florida Cancer Specialists and Research Institute - Panhandle Region, Tallahassee, Florida
  - Florida Cancer Specialists and Research Institute, West Palm Beach, Florida
  - University Cancer and Blood Center, Athens, Georgia
  - Cancer Treatment Centers of America, Newnan, Georgia
  - University of Chicago Medical Center - Duchossois Center for Advanced Medicine (DCAM), Chicago, Illinois
  - Orchard Healthcare Research, Skokie, Illinois
  - American Health Network, Indianapolis, Indiana
  - Baptist Health Lexington, Lexington, Kentucky
  - SMHC Cancer Care and Blood Disorders, Biddeford, Maine
  - University of Maryland - Greenebaum Comprehensive Cancer Center, Baltimore, Maryland
  - GBMC Cancer Center, Baltimore, Maryland
  - Chevy Chase Health Care Center/ RCCA, Chevy Chase, Maryland
  - James M. Stockman Cancer Institute, Frederick, Maryland
  - Maryland Oncology Hematology, P.A., Rockville, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Cancer and Hematology Centers of Western Michigan, Grand Rapids, Michigan
  - Virginia Piper Cancer Institute, Allina Health, Minneapolis, Minnesota
  - Forrest General Cancer Center/Hattiesburg Clinic, Hattiesburg, Mississippi
  - Jackson Oncology Associates, Jackson, Mississippi
  - Mercy Cancer Center, Joplin, Missouri
  - HCA Midwest Health, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital St. Louis, David C. Pratt Cancer Center, St Louis, Missouri
  - St. Vincent Frontier Cancer Center, Billings, Montana
  - Oncology Hematology West, P.C. dba Nebraska Cancer Specialists, Papillion, Nebraska
  - New Jersey Hematology Oncology Associates, Brick, New Jersey
  - Regional Cancer Care Associates, East Brunswick, New Jersey
  - The Valley Hospital, Ridgewood, New Jersey
  - Regional Cancer Care Associates, LLC-Sparta, Sparta, New Jersey
  - New Mexico Cancer Care Alliance - Southwest Gynecology Oncology, Albuquerque, New Mexico
  - New York Oncology Hematology, P.C., Albany, New York
  - New York Cancer and Blood Specialists, East Setauket, New York
  - Hematology Oncology Associates of Central New York, P.C., East Syracuse, New York
  - Broome Oncology, LLC, Johnson City, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of North Carolina Lineberger Cancer Center, Chapel Hill, North Carolina
  - Ohio State University Comprehensive Cancer Center, Stephanie Spielman Comprehensive Breast Center, Columbus, Ohio
  - Mercy Clinic Oncology and Hematology, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute, LLC, Tulsa, Oklahoma
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - Cancer Treatment Centers of America - Philadelphia, Philadelphia, Pennsylvania
  - Magee-Women's Hospital of UPMC, Pittsburgh, Pennsylvania
  - West Cancer Center, Germantown, Tennessee
  - Sarah Cannon Research Institute at Tennessee Oncology, Nashville, Tennessee
  - Texas Oncology - Bedford, Bedford, Texas
  - Texas Oncology - Medical City Dallas, Dallas, Texas
  - Texas Oncology - Dallas Presbyterian Hospital, Dallas, Texas
  - Texas Oncology - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Texas Oncology - Memorial City, Houston, Texas
  - Westside Surgical Hospital and Breast Center, Houston, Texas
  - Oncology Consultants, Houston, Texas
  - Hope Cancer Center of East Texas, Tyler, Texas
  - Bon Secours St. Francis, Midlothian, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - Overlake Medical Center, Bellevue, Washington
  - Kadlec Regional Medical Center, Kennewick, Washington
  - Swedish Cancer Center, Seattle, Washington
  - Northwest Medical Specialties, Tacoma, Washington
- Australia (9):
  - Border Medical Oncology, Albury, New South Wales
  - Sydney Adventist Hospital, Wahroonga, New South Wales
  - Mater Cancer Care Centre, South Brisbane, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Monash Medical Centre, Clayton, Victoria
  - Peninsula and South Eastern Haematology and Oncology Group, Frankston, Victoria
  - Breast Cancer Research Centre, Nedlands, Western Australia
  - St. John of God Subiaco Hospital, Perth, Western Australia
  - Flinders Medical Centre, Bedford Park
- Austria (4):
  - Universitätsklinik Onkologie Landeskkrankenhaus, Salzburg
  - Facharzt für Frauenheilkunde und Geburtshilfe Spezialist für Brustchirurgie und Brustkrebs, Schwaz
  - Ludwig Boltzmann Institut fur Klinische Onkologie und Photodynamische Therapie, Vienna
  - AKH-Frauenheilkunde, Vienna
- Belgium (5):
  - AZ Klina AUGUSTIJNSLEI, Antwerp
  - Institut Jules Bordet, Brussels
  - UZA, Edegem
  - UZ Leuven, Leuven
  - CHC-Sant Joseph Oncology-Hematology, Liège
- Canada (9):
  - The Moncton Hospital, Moncton, New Brunswick
  - QEII Health Sciences Centre - Nova Scotia Cancer Centre, Halifax, Nova Scotia
  - St. Michael's Hospital, Toronto, Ontario
  - Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - Center Hospitalier de Montreal CHUM McPeak Sirois, Montreal, Quebec
  - CIUSSS de Centre-Ouest-de-l'Île-de-Montréal Jewish General Hospital, Montreal, Quebec
  - McGill University Health Center, Montreal, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke CIUSSS de lEstrie CHUS patyre, Sherbrooke, Quebec
  - CHU de Quebec-University Laval, Québec
- Czechia (4):
  - NH Hospital a.s. Nemocnice Hořovice Onkologie, Hořovice
  - Onkologicka Klinika FN Olomouc, Olomouc
  - Onkologicka Klinika (Vseobecna Fakultni Nemocnici v Praze ), Prague
  - Onkologicka Klinika (Fakultni Nemocnice v Motole), Prague
- France (7):
  - CHRU J. Minjoz Service Oncologie, Besançon
  - Centre François Baclesse Service the Recherche Clinique, Caen
  - Hospices Civils de Lyon Sud Oncologie Medicale, Pierre-Bénite
  - Centre Eugène Marquis, Rennes
  - Institut Curie - Hopital Rene Huguenin, Saint-Cloud
  - Clinique Sainte Anne - Strasbourg Oncologie Liberale, Strasbourg
  - Centre Hospitalier Regional et Universitaire de Tours CHRU, Tours
- Germany (11):
  - St. Elisabeth-Krankenhaus GmbH, Cologne, North Rhine-Westphalia
  - InVO - Institut für Versorgungsforschung, Koblenz, Rhineland-Palatinate
  - St. Elisabethgruppe GmbH Marien Hospital Witten Brustzentrum, Witten, Rhineland-Palatinate
  - Arzt der Studienzentrale Universitätsklinikum Erlangen, Erlangen, State of Berlin
  - Charité Universitätsmedizin Berlin-Campus Benjamin Franklin Klinik für Hämatologie, Onkologie und Tumorimmunologie, Berlin
  - Helios Klinikum Berlin-Buch, Berlin
  - Mammazentrum HH am Krankenhaus Jerusalem, Hamburg
  - UKSH, Campus Kiel Klinik für Gynäkologie und Geburtshilfe, Kiel
  - Staedtisches Klinikum Lueneburg gGmbH Brustzentrum und gynaekologisches Krebszentrum der Frauenklinik, Lüneburg
  - LMU Klinikum der Universität München Breast Cancer, München
  - Technische Universität München Klinikum rechts der Isar Klinik und Poliklinik für Frauenheilkunde, München
- Hungary (6):
  - Military Hospital State Health Center, Budapest
  - Országos Onkológiai Intézet, Budapest
  - Semmelweis University, Budapest
  - Uzsoki utcai kórház, Budapest
  - Szabolcs Szatmar Bereg Megyei Korhazak Es Egyetemi Oktatokorhaz, Nyíregyháza
  - University of Pécs Department of Oncotherapy, Pécs
- Italy (4):
  - Ospedale San Raffaele - Medical Oncology Dept., Milan
  - Istituto Europeo di Oncologia (IEO), Milan
  - Centro Oncologico Modenese, Modena
  - S.C. Oncologia/Az. Osp.Ra. S Maria Terni, Terni
- Poland (6):
  - Szpitale Pomorskie Oddział Onkologii i Radioterapii Powstania, Gdynia
  - Samodzielny Publiczny Zespol Gruzlicy i Chorob Pluc, Oddzial Onkologii z Pododdzialem Chemoioterapii, Olsztyn
  - Mrukmed, Rzeszów
  - Klinika Nowotworów Piersi i Chirurgii Rekonstrukcyjnej Centrum Onkologii-Instytut, Warsaw
  - Wilmed, Warsaw
  - Onko-Dent G.L.Slomian, Żory
- Russia (2):
  - State Oncology Clinical Dispansery, Saint Petersburg
  - Federal State Budgetary Institution Research Institute of Oncology named after N.N. Petrov of the Ministry of Health of the Russian Federation, Saint Petersburg
- Singapore (3):
  - John Hopkins Singapore International Medical Centre, Singapore
  - National Cancer Centre Singapore, Singapore
  - National University Hospital, Singapore
- South Korea (11):
  - Dong-A University Hospital, Busan
  - Kyungpook National University Hospital, Daegu
  - National Cancer Center, Goyang
  - Gachon University Gil Medical Center, Incheon
  - Gangnam Severance Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Ajou University Hospital, Suwon
  - St. Vincents Hospital, Suwon
- Spain (14):
  - Onkologikoa, San Sebastián, Gipuzkoa
  - Althaia Hospital Sant Joan de Deu, Barcelona, Manresa
  - Hospital Teresa Herrera Materno-Infantil (CHUAC), A Coruña
  - Centro Oncológico de Galicia, A Coruña
  - Hospital Quironsalud Barcelona, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Institut Catala d'Oncologia, Barcelona
  - HU San Pedro de Alcantara, Cáceres
  - Hospital Universitario Ramon y Cajal Servicio de Oncologia, Madrid
  - IOB_Hospital Ruber Internacional, Madrid
  - Fundacion Jimenez Diaz, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Miguel Servet Paseo Isabel la Catolica 1-3 Edificio de Maternidad, Zaragoza
- Taiwan (7):
  - Changhua Christian Hospital, Taichung
  - Chi Mei Medical Center, Tainan
  - National Cheng Kung University Hospital, Tainan
  - Koo Foundation Sun Yat-Sen Cancer Center, Taipei
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital Linkou Branch, Taoyuan District
- Thailand (3):
  - Chulabhorn Hospital, Bangkok
  - King Chulalongkorn Memorial Hospital, Bangkok
  - Buddhachinaraj Hospital, Phitsanulok
- Ukraine (8):
  - Dnipropetrovsk City Multifield Clinical Hospital #4, Dnipro
  - Communal Non-Profit Enterprise "Regional Center of Oncology", Kharkiv
  - Kryviy Rih Onkology Dispensary, Kryvyi Rih
  - National Cancer Institute, Kyiv
  - Municipal Institution of Lviv Regional Council - Lviv Oncology Regional Treatment Diagnostic Center, Lviv
  - Central City Clinical Hospital, City Oncology Center, Uzhhorod
  - Podilskiy Regional Center of Oncology, Vinnytsia
  - Communal Institution "Zaporizhzhia Regional Clinical Oncological Dispensary", Zaporizhzhia
- United Kingdom (4):
  - Royal Cornwall Hospital Oncology Trials, Sunrise Centre, Truro, Cornwall
  - Hertford County Hospital, Hertford
  - Cancer Centre, Guy's Hospital, London
  - Nottingham University Hospitals NHS Trust, Nottingham

IPD SHARING:
Plan to Share IPD: Undecided
Currently under evaluation by the organization